CLINICAL TRIAL: NCT07095465
Title: 52-Week, Phase 3, Open-Label Extension Study of ACP-204 in Adults With Lewy Body Dementia Psychosis (LBDP)
Brief Title: Phase 3, Open Label Extension Study of ACP-204 in Lewy Body Dementia Psychosis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-204-013; 2025-521711-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-07

CONDITIONS: Lewy Body Dementia Psychosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACP-204 (Experimental): Initiation of treatment with ACP-204 at a dose of 30 mg once daily. During the trial, the dose may be adjusted, i.e. uptitration to 60 mg in case of suboptimal efficacy or subsequent down titration to 30 mg. Repeated titration steps are allowed.
  Interventions: Drug: ACP-204

INTERVENTIONS:
Drug: ACP-204 — Provided as 1 capsule, to be taken orally once daily
  Other Names: ACP-204 Tartrate

SUMMARY:
A 52-Week, Phase 3, Open-Label Extension Study of ACP-204 in Adults With Lewy Body Dementia Psychosis (LBDP)

ELIGIBILITY:
Inclusion Criteria:

* The subject may benefit from long-term therapy with open-label ACP-204 treatment in the judgment of the Investigator
* Subject has completed Visit 6 (EOT) of the antecedent ACP-204-012 study and did not have an early discontinuation from the antecedent study
* Can complete all study visits with a study partner/caregiver
* Can understand the nature of the study and protocol requirements and provide written informed consent. If the subject is deemed not competent to provide informed consent, the following requirements for consent must be met:

  1. The subject's LAR (or study partner/caregiver, if local regulations allow) must provide written informed consent.
  2. The subject must provide written (if capable) informed assent per local regulations
* If the subject is a female, she must be of nonchildbearing potential
* If the subject is male, he must agree to the following during the study intervention period and for at least 90 days after the last dose of study drug:

  1. Refrain from donating sperm, AND
  2. Either

     * Be abstinent from sexual intercourse where pregnancy can occur (abstinent on a long-term and persistent basis) and agree to remain abstinent OR
     * Use a condom and subject's female partner (if of childbearing potential and not pregnant) must use an additional contraceptive method

Exclusion Criteria:

* Is judged by the Investigator or the Medical Monitor to be inappropriate for the study for any reason
* Is in hospice, is receiving end-of-life palliative care, or is bedridden
* Has a heart rate <50 beats per minute, as measured by vital signs at Baseline (EOT visit of the antecedent study). If bradycardia is secondary to iatrogenic or treatable causes and these causes are addressed, a heart rate assessment can be repeated.
* Has a BMI <18.5 kg/m2 or known unintentional weight loss ≥7% of body weight over past 6 months
* Has a clinically significant laboratory abnormality in the antecedent ACP-204-012 study, excepting at ACP-204-012 EOT, that in the judgment of the Investigator or Medical Monitor, will either:

  1. jeopardize the safe participation of the subject in this study; OR
  2. interfere with the conduct or interpretation of safety or efficacy evaluations in the study
* Is actively suicidal at Visit 1 (Baseline, EOT visit of the antecedent study)
* Has a neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical or mental disorder, including cancer or malignancies that, in the judgment of the Investigator, would increase the risk associated with taking study medication or significantly interfere with the conduct or interpretation of the study
* Requires treatment with a medication or other substance that is prohibited by the protocol or will be used in a way that violates a use restriction

Ages: 55 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who experience treatment-emergent adverse events (TEAEs) | 52 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Humanity Clinical Research, Corp, Aventura, Florida
  - K2 Summit Research, Lady Lake, Florida
  - Homestead Associates in Research Inc, Miami, Florida
  - Advanced Clinical Research Network, Corp, Miami, Florida
  - Health Synergy Clinical Research, LLC, West Palm Beach, Florida
  - R and H Clinical Research, Stafford, Texas

IPD SHARING:
Plan to Share IPD: No